CLINICAL TRIAL: NCT00922025
Title: A Multi-centre, Naturalistic Study to Explore the Correlation Between Smoking Pattern and Clinical Efficacy of EGFR TKI in Male Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer of Adeno Histology Failed 1st Line Chemotherapy
Brief Title: Multicentre Study to Explore the Correlation Between Smoking Pattern and Clinical Efficacy of Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor (TKI) in Male Patients
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OTW-IRE-2009/1
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; Male; Smoking Pattern; Efficacy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Male patients with non-small cell lung cancer (NSCLC) of adeno histology

SUMMARY:
The objective is to investigate the correlation between smoking pattern and clinical efficacy of EGFR TKIs in male patients with locally advanced or metastasized non-small cell lung cancer of adeno histology who have failed 1st line chemotherapy. Health care resource usage, quality of life (EQ-5D) and practice of EGFR mutation test will also be evaluated. Current practice of EGFR mutation testing in Taiwan will be surveyed.

ELIGIBILITY:
Inclusion Criteria:

* Male patients age 20 years or older
* Histological or cytological confirmation of NSCLC of adeno histology. If sputum is the only available sample, a second positive test is necessary for cytological confirmation
* Locally advanced or metastatic on or after first-line chemotherapy. Imaging evidence of disease progression can be either chest X ray, CT or MRI assessment on measurable lesions. If no measurable lesion is available, evaluable lesions are acceptable

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2009-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Correlation between smoking patterns and best objective tumor response rate | 6 Months

SECONDARY OUTCOMES:
correlation between smoking patterns and progression free survival (PFS) | 9 months
correlation between smoking patterns and overall survival (OS) | 9 Months
changes from baseline in quality of life questionnaires (EQ-5D) after EGFR-TKI therapy | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Ming Tsai, MD, Principal Investigator — Taipei Ventrans General Hospital
Locations (6):
- Taiwan (6):
  - Research Site, Changhua
  - Research Site, Chiayi City
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei